CLINICAL TRIAL: NCT00774787
Title: A Randomized, Open-label, Assessor-blinded, Split-face Study of Imiquimod 5% Cream Applied After Cryotherapy of Actinic Keratoses
Brief Title: Topical Imiquimod Cream in Combination With Cryotherapy for the Treatment of Actinic Keratoses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigel Dermatology (Other)
Responsible Party: Principal Investigator, Darrell S. Rigel, PI, Rigel Dermatology
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 08US02IMIQ-Rigel
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Results first posted 2010-10-27 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-10

CONDITIONS: Actinic Keratoses
Keywords: Combination treatment; Imiquimod; Cryotherapy
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imiquimod, treatment, topical cream (Experimental): Imiquimod 5% cream, 1 packet (250 mg cream), applied to left or right treatment area on the face and/or balding scalp
  Interventions: Drug: imiquimod 5% cream
- Control, Untreated (No Intervention): No treatment of treatment area on the other half of the face and/or balding scalp

INTERVENTIONS:
Drug: imiquimod 5% cream — 1 packet (250 mg cream) 3 times per week for 4 weeks
  Other Names: Aldara
  Arms: Imiquimod, treatment, topical cream

SUMMARY:
The purpose of this study is to determine if use of topical imiquimod cream after cryotherapy of actinic keratoses reduces the total number of lesions (those treated with cryotherapy and new ones) at follow-up.

DETAILED DESCRIPTION:
Actinic keratoses are common skin lesions associated with excess sun exposure. Over time, there is a small risk a lesion may progress to skin cancer. Since one can not predict which actinic keratosis will progress, the standard of care is to treat the lesions. The most commonly used method to treat actinic keratoses in the United States is with cryotherapy, which uses intense cold to freeze and destroy the lesions. Efficacy appears to be related to how long one freezes the lesion, but increasing the freeze time may result in increased pain and/or skin pigment changes after treatment.

Cryotherapy is a provider-administered "focal" treatment that only treats the lesions that are frozen. There may be early actinic keratoses in the skin surrounding treated lesions that are not easily seen; these may progress over time to visible lesions. There several patient-administered topical treatments for actinic keratoses that are applied to a treatment area or "field" rather than to specific lesions. Imiquimod 5% cream is one such treatment, and is approved in the United States for the treatment of AKs with a dosing regimen of 1 packet applied 2 times per week to a 25 cm2 area 2x/week for 16 weeks.

The study will use a split-face design (one side of face treated and the other side untreated) to explore whether a 4-week course of topical imiquimod 5% cream after cryotherapy of actinic keratoses reduces the total number of lesions (those treated with cryotherapy and new ones) in the treatment area at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of actinic keratoses
* Actinic keratoses in two reasonably bilaterally symmetric areas on the face and/or balding scalp:

  * each area with a minimum of 25 cm^2 and a maximum of 50 cm^2
  * each area with at least 6 typical, non-hypertrophic target AKs
  * with target AK lesion counts of +/- 1 lesion between the areas
  * each area that the patient can distinguish with respect to study drug application
* Able to comply with all study requirements
* Are willing and able to give written informed consent

Exclusion Criteria:

* Uncontrolled intercurrent or chronic illness
* Systemic immunocompromise due to disease or treatment
* Clinically relevant systemic autoimmune disease
* Pregnant or nursing
* Dermatologic disease and/or condition in the treatment area that may be exacerbated by imiquimod or cause difficulty with examination
* Participation in another clinical study
* Allergies to imiquimod or any of the excipients in the cream
* Treatment within the past 90 days with any of the following:

  * Psoralens plus ultraviolet A therapy
  * Ultraviolet B therapy
  * Systemic immunomodulators (e.g. oral or parenteral corticosteroids at greater than physiologic doses, interferons, anti-TNF agents, cytokines)
  * Chemotherapeutic or cytotoxic agents;
  * Investigational agent
* Treatment within the past 30 days with any of the following:

  * Surgical excision
  * Photodynamic therapy
  * Curettage
  * Topical corticosteroids
  * Laser
  * Dermabrasion
  * Chemical peel
  * Imiquimod 5% cream
  * Topical retinoids
  * 5-fluorouracil
  * Masoprocol
  * Pimecrolimus or tacrolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darrell S Rigel, MD, Study Chair — Rigel Dermatology; James Q Del Rosso, DO, Principal Investigator — Private Practice; James Spencer, Principal Investigator — Spencer Dermatology
Locations (3):
- United States (3):
  - Spencer Dermatology and Skin Surgery, St. Petersburg, Florida
  - James Del Rosso, Henderson, Nevada
  - Rigel Dermatology, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled - 08 Oct 08; last patient enrolled - 07 Jul 09; last patient completed: 09 Sep 09; Setting - private practice clinics
Groups:
- Cryotherapy Followed by Imiquimod 5% Cream or Observation: Split-face study of cryotherapy of all actinic keratoses in target treatment area (bilaterally symmetrical area on face or balding scalp) followed by random assignment to treatment of half of treatment area with imiquimod 5% cream and of other half to no treatment
Period: Overall Study
Arm/Group | Cryotherapy Followed by Imiquimod 5% Cream or Observation
Started | 27
Completed | 26
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cryotherapy Followed by Imiquimod 5% Cream or Observation
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 27
Actinic keratoses, total [Mean (Standard Deviation); unit: Lesions] — Total count of clinically diagnosed actinic keratoses in target treatment area
  Lesions | 17.3 (4.1)
Actinic keratoses, Imiquimod side [Mean (Standard Deviation); unit: Lesions] — Count of actinic keratoses on side of target treatment area randomly assigned to imiquimod 5% cream following cryotherapy
  Lesions | 8.7 (2.2)
Actinic keratoses, Observation Side [Mean (Standard Deviation); unit: Lesions] — Count of actinic keratoses on side of target treatment area randomly assigned to observation following cryotherapy
  Lesions | 8.5 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Actinic Keratoses Count at 4-8 Weeks Post-treatment
Description: Percent change = [(actinic keratoses count at 4-8 weeks post-treatment)-(actinic keratoses count at baseline)]/(actinic keratoses count at baseline)]*100%. Data from one patient, lost to follow-up immediately after cryotherapy, not included in these analyses. Actinic keratoses at 4-8 weeks post-treatment visit includes all actinic keratoses in each respective treatment area, baseline and new.
Time Frame: Baseline, 4-8 weeks post-treatment
Population: Patients who had end of study visit with count of actinic keratoses. Change not calculated for one patient who was lost to follow-up immediately after baseline visit, and had no post-treatment data. Actinic keratoses at 4-8 weeks post-treatment visit includes all actinic keratoses in each respective treatment area, baseline or new.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cryotherapy Followed by Imiquimod 5% Cream or Observation
Number analyzed (Participants) | 26
Percent change
  Change from baseline, imiquimod side | -73.2 (27.1)
  Change from baseline, observation side | -62.0 (30.3)

2. Post Hoc Outcome: Complete Clearance of Actinic Keratoses at 4-8 Weeks Post-treatment
Description: Complete clearance (actinic keratosis count of 0) in each respective area at 4-8 weeks post-treatment. Actinic keratoses at 4-8 weeks post-treatment visit includes all actinic keratoses in each respective treatment area, baseline and new.
Time Frame: 4-8 weeks post-treatment
Population: All patients enrolled.
Measure: Number; unit: Participants
Units Other Than Participants: Treatment areas
Arm/Group | Cryotherapy Followed by Imiquimod 5% Cream or Observation
Number analyzed (Participants) | 27
Number analyzed (Treatment areas) | 27
Participants
  Completely cleared, imiquimod side | 8
  Completely cleared, observation side | 5

3. Secondary Outcome: Cosmetic Appearance Score at 4-8 Weeks Post-treatment
Description: Cosmetic appearance score, based recall comparison to appearance at baseline. Seven point scale: +3 = treatment area is much better appearing; +2 = treatment area is moderately better appearing; + 1 = treatment area is slightly better appearing; 0 = treatment area appears same; -1 = treatment area is slightly worse appearing; -2 = treatment area is moderately worse appearing; -3 = treatment area is much worse appearing. Data from one patient, lost to follow-up immediately after cryotherapy, not included in these analyses.
Time Frame: 4-8 weeks post-treatment
Population: Patients who had end of study visit with cosmetic appearance assessment. Cosmetic appearance score, by treatment area, not included for one patient who was lost to follow-up immediately after baseline visit, and had no post-treatment data.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cryotherapy Followed by Imiquimod 5% Cream or Observation
Number analyzed (Participants) | 26
Scores on a scale
  Investigator assessed, imiquimod side | 2.1 (1.1)
  Investigator assessed, observation side | 1.6 (1.1)
  Patient assessed, imiquimod side | 2.6 (1.0)
  Patient assessed, observation side | 1.2 (1.3)

4. Other Pre Specified Outcome: Local Skin Reactions
Description: Mean maximum post-baseline intensity of investigator assessed local skin reactions (erythema, edema, weeping/exudate, flaking/scaling/dryness, scabbing/crusting, erosion/ulceration) by treatment area. 0 = none, 1 = mild, 2 = moderate, 3 = severe. Data from one patient, lost to follow-up immediately after cryotherapy, not included in these analyses.
Time Frame: Post baseline to end of study (4-8 weeks post-treatment)
Population: One patient not included who was lost to follow-up immediately after baseline visit, and had no post-treatment data.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cryotherapy Followed by Imiquimod 5% Cream or Observation
Number analyzed (Participants) | 26
Scores on a scale
  Erythema, imiquimod side | 1.5 (0.7)
  Erythema, observation side | 1.3 (0.5)
  Edema, imiquimod side | 0.2 (0.4)
  Edema, observation side | 0.1 (0.3)
  Weeping/exudate, imiquimod side | 0.3 (0.7)
  Weeping/exudate, observation side | 0.0 (0.0)
  Flaking/scaling/dryness, imiquimod side | 1.4 (0.6)
  Flaking/scaling/dryness, observation side | 1.2 (0.6)
  Scabbing/crusting, imiquimod side | 0.9 (1.1)
  Scabbing/crusting, observation side | 0.6 (0.7)
  Erosion/ulceration, imiquimod side | 0.4 (0.7)
  Erosion/ulceration, observation side | 0.1 (0.4)

ADVERSE EVENTS:
Time Frame: 8-12 weeks: from baseline cryotherapy visit to end of study (4-8 weeks post completion of imiquimod treatment).
Arm/Group | Cryotherapy Followed by Imiquimod 5% Cream or Observation
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 3/27
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryotherapy Followed by Imiquimod 5% Cream or Observation (N=27)
Systemic interferon reaction on areas with previous sun exposure; arms, thighs, upper chest, upper b (Skin and subcutaneous tissue disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Decreased appetite (Gastrointestinal disorders) | 1 (1)
Cold (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Open label; small patient number; planned secondary endpoint of change in only lesions treated with cryotherapy (baseline) not determinable as only all lesions (baseline + new) consistently captured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs must agree on communication of complete results, but may discuss individual site results. Collaborator can review complete results communications prior to public release and can embargo communications regarding trial results, if patents are to be pursued, for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the collaborator for review. The collaborator cannot require changes to the communication and cannot extend the embargo.